CLINICAL TRIAL: NCT03271775
Title: Vestibulopathy With Vestibulo Ocular Reflex (VOR) Gain Deficit - Characteristics of Overt and Covert Saccadic Eye Movements Measured by the Video Head Impulse Test (vHIT)
Brief Title: Vestibulopathy With Vestibulo Ocular Reflex (VOR) Gain Deficit
Acronym: VOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Carmeli Eli, Prof., University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHaifa2808
Record Dates: First submitted 2017-08-02; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Vestibulopathy, Acute Peripheral
Keywords: Dizziness; Instability
MeSH Terms: conditions — Vestibular Neuronitis; Dizziness | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: After the initial test, subjects will randomly distribute into three different research groups.
  Each subgroup will include 30 patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Patients in the control group will follow the doctor's instructions (medications and etc.) and will not participate in any physical therapy program.
- PT treatment group for balance disorder (Experimental): Patients in this research group will join to a 3 months' physical therapy treatment group designed to improve balance. The service for the group is provided by laboratory.
  Interventions: Other: physical therapy program (group)
- independant home computerized exercises (Experimental): Patients in this group will be treated by 3 months' independent home computerized exercise program. Each patient will receive a personal access code for the exercise program. The duration of each practice is 5-10 minutes per day.
  Interventions: Other: physical therapy program (computerized exercises)

INTERVENTIONS:
Other: physical therapy program (group) — Exercises group transmitted by physical therapist (Up to four participant in each group).
  Arms: PT treatment group for balance disorder
Other: physical therapy program (computerized exercises) — Remote exercises program accompanied by a physical therapist guidance
  Arms: independant home computerized exercises

SUMMARY:
The study is examine the eye movements characteristics of patients with VOR gain deficits (overt and covert saccades) before and after physical therapy intervention program and examine the most effective physical therapy treatment program for patients with vestibulopathy.

DETAILED DESCRIPTION:
The vestibular system receives and conveys information about head motion in space, and is the main human sensory system dedicated to detecting self-motion.The vestibular system plays a crucial role in static and dynamic balance control, stabilizing the head and trunk, especially on unstable surfaces . In terms of postural control and falls, the literature describes a direct association between VOR deficits, gait instability, and falls.The "gain" of the VOR is defined as the change in the eye angle divided by the change in the head angle during the head turn. Under ideal conditions, the gain of the rotational VOR is 1.0, meaning there is a compensatory eye velocity equal to the head velocity and in the opposite direction. In case of a positive vHIT, the VOR gain is decreased and refixating saccades are observed. The video Head Impulse Test measures eye velocity during head rotation. Instant feedback about every single head impulse allows the examiner to apply a set of standardized graded impulses. The system is easy to use in a clinical setting, provides an objective measure of the VOR, and detects both overt and covert catch-up saccades in patients with vestibular loss. Measurements are quick and noninvasive, and the automated analysis software provides instant results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral or bilateral vestibulopathy living independently in the community

Exclusion Criteria:

* cognitive state decline neurological disorder disease or disorders that can affect balance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline saccadic eye movements after 3 and 6 months measured by The video head impulse test (vhit) | up to 7 days after acute vestibulopathy, after 3 and 6 months after acute vestibulopathy
  The Vhit incorporates a new technology that uses a high speed light weight video goggle to measure high velocity and record "catch up" saccades in patients with impaired VOR function. we will examine the changes from baseline in the latency, frequency and duration of the overt and covert saccadic eye movements. In addition, we would like to examine changes over time in the ratio between the head and the eye movement (Gain).

SECONDARY OUTCOMES:
Change from baseline velocity sway at 3 and 6 months measured by force platform | up to 7 days after acute vestibulopathy, after 3 and 6 months after acute vestibulopathy
  The force plate is designed to measure the forces and moments applied to its top surface as a subjects stands, steps, or jumps on it. Force plates are regularly used in research and clinical studies looking at balance, gait, and sports performance (www.amti.biz). Center of pressure (COP) data during the stability tests will be sampled at a frequency of 100 Hz. We will perform the zur balance scale (ZBS) on the plate at each time and evaluate the changes from baseline.
Changes from baseline in balance confidence at 3 and 6 months after vestibulopathy measured by the ABC questionnire | up to 7 days after acute vestibulopathy, after 3 and 6 months after acute vestibulopathy
  The ABC is one of a several tools designed to measure an individual's confidence in her/his ability to perform daily activities without falling.

CONTACTS AND LOCATIONS:
Overall Officials: Carmeli Eli, Prof, Principal Investigator — Haifa University
Locations (1):
- Israeli Center for the Treatment of Dizziness and Imbalance, Raanana, Israel

IPD SHARING:
Plan to Share IPD: Yes
the data for all primary and secondary outcome measure will be available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: data will be available within 6 months of study completion
Access Criteria: Requestor will be required to sign a data access agreement